CLINICAL TRIAL: NCT06134791
Title: Differences in Headache Characteristics of a Subgroup of Cervicogenic Headache Patients With a Positive or Negative FRT: a Cross-sectional Comparison.
Brief Title: Differences in Characteristics of Headache Patients With a Positive or Negative FRT: a Cross-sectional Comparison.
Status: Recruiting | Type: Observational
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: BC-10474 AM2
Record Dates: First submitted 2023-07-06; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Headache
MeSH Terms: conditions — Headache

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cervicogenic headache with positive flexion-rotation test: Diagnosis of cervicogenic headache according to the ICHD-3 criteria. Age: 18+ years Headache for at least 1 day/week for at least 3 months Limited mobility of the neck Positive flexion-rotation test (<32 degrees on the left/right side or a difference of 10 degrees or more between left and right side) NPRS > 3/10
  Interventions: Other: No intervention
- Cervicogenic headache without positive flexion-rotation test: Diagnosis of cervicogenic headache according to the ICHD-3 criteria Age: 18+ years Headache for at least 1 day/week for at least 3 months Limited mobility of the neck Negative flexion-rotation test (>32 degrees on the left/right side or a difference of less than 10 degrees between left and right side) NPRS > 3/10
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
An observational study will be conducted to evaluate the differences in headache characteristics between a subgroup of cervicogenic headache patients with a positive and negative flexion-rotation test at the C1-C2 level. Differences may guide future treatment allocation and the use of more individualized treatment options.

DETAILED DESCRIPTION:
Headache is a common and disabling condition. Several primary and secondary headache forms have been described, such as migraine, tension-type headache and cervicogenic headache (CH). In patients with CH; we can see a referred pain pattern to the head, possibly originating from a source in the (upper)cervical spine. It has been described that nociceptive input, originating from the C1-C3 nervous system may be responsible for pain referral to head and neck regions. Recently, the flexion-rotation test (FRT) has been described as one of the most useful clinical tests in the clinical testing and research of CH. Other literature showed that the rotational movement during the FRT was diminished in patients with CH and these results were correlated to headache intensity.

To treat this disabling condition, manual therapy is already known to be an effective treatment strategy. However, the additional value of dry needling is still to be discussed. Since the M. Obliquus capitis inferior (M. OCI) finds its origin on the apex of the spinous processus of C2 and inserts on transverse processus of the atlas (C1); this muscle might be anatomically very relevant to influence rotational mobility in the upper cervical spine. Additionally, this muscle is responsible for proprioception and accurate positioning of the head and neck, due to the presence of a large amount of Golgi bodies and muscle spindles in the muscle. Considering the myofascial pain referral pattern of the M. OCI, a referred pain pattern to the temporal region may be present when active triggerpoints are present.

Previous research already showed some preliminary evidence for positive treatment effects by dry needling of the M. OCI in patients with cervicogenic dizziness and headache.

The goal of this study is to evaluate the differences in headache characteristics between a subgroup of cervicogenic headache patients with a positive and negative flexion-rotation test at the C1C2 level. Differences may guide future treatment allocation and the use of more individualized treatment options.

In this observational study, 100 patients with cervicogenic headache will be recruited. Participants are required to have complaints for at least 3 months. Participants are included based on online questionnaires and a clinical examination of the neck and shoulder region. All participants will receive information and have to sign an informed consent form.

Participants will be subjected to a single assessment, which involves questionnaires and measurements of the cervical spine.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cervicogenic headache according to the ICHD-3 criteria:

A. Any headache fulfilling criterion C B. Clinical and/or imaging evidence1 of a disorder or lesion within the cervical spine or soft tissues of the neck, known to be able to cause headache2

C. Evidence of causation demonstrated by at least two of the following:

* headache has developed in temporal relation to the onset of the cervical disorder or appearance of the lesion
* headache has significantly improved or resolved in parallel with improvement in or resolution of the cervical disorder or lesion
* cervical range of motion is reduced, and headache is made significantly worse by provocative manœuvres
* headache is abolished following diagnostic blockade of a cervical structure or its nerve supply D. Not better accounted for by another ICHD-3 diagnosis

Age: 18+ years Headache for at least 1 day/week for at least 3 months Limited mobility of the neck NPRS > 3/10

Exclusion Criteria:

* Primary headache forms: migraine, TTH
* Other secondary headaches that do not comply with the ICDH-3 criteria for CH
* Whiplash or other traumatic incident in the past
* Pregnancy or given birth in the last year
* Previous head, neck or shoulder surgery
* Cervical radiculopathy complaints
* Receiving other treatments for headache or neck pain (physical therapy/ostheopathy/chiropraxie...) in the previous month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with chronic headache, compliant to the ICHD-3 criteria for cervicogenic headache.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Headache pain intensity | Baseline
  Subjects will have to report their actual pain complaints on a numeric pain rating scale (NPRS) ranging from 0 (no pain) to 10 (worst pain) at baseline testing.
Headache frequency | Baseline
  Frequency of headache attacks will be registered
Headache duration | Baseline
  Duration of headache attacks will be registered
Headache related disability | Baseline
  Headache related disability will be questioned using the Henry Ford Headache Disability Index (HDI). The total score ranges from 0-100. The higher the score, the more disabilitating the headache is for the patient.
Headache related impact | Baseline
  Headache related disability will be questioned using the Headache Impact Test (HIT-6) questionnaire. The total score can range from 36 to 78, with a higher score indicating the headache has more impact on daily life.
Neck pain intensity | Baseline
  Subjects will have to report their actual pain complaints on a numeric pain rating scale (NPRS) ranging from 0 (no pain) to 10 (worst pain) at baseline testing.
Neck disability | Baseline
  Neck pain related disability will be questioned using the NDI (Neck Disability Index). The total score ranges from 0 to 50, with a higher score indicating more disability.

SECONDARY OUTCOMES:
Pain Pressure Thresholds (PPTs) | Baseline
  PPT measurements will be registered with the digital hand-held pressure algometer (Wagner FPX 25 Force Gage).
  To standardize the pressure applied by the investigator, the same investigator always stabilized his wrist with his other hand. The PPT assessment was performed two times with a 30-second break between each application and the pressure will be increased by 1N/s until the patient reports the pressure as unpleasant. This pressure will be taken as PPT expressed in Newton (N); and the average will be taken of the three measurements on the spinous process of C2 and the Upper Trapezius Muscle (bilateral measurement).
Joint Position Error | Baseline
  Joint position error will be registered with the digital Motion Guidance Laser.
  The Cervical Joint Position Error (JPE) Test is a measurement tool used to clinically assess an individual's cervicocephalic proprioception ability. Cervicocephalic proprioception describes one's sense of position of their head and neck in space. The Cervical JPE Test measures the ability of a blindfolded patient to accurately relocate their head position back to a predetermined neutral point after cervical joint movement. The average of 6 measurements to each side will be used to determine JPE.
Global active range of motion of the cervical spine. | Baseline
  Changes in global cervical mobility will be assessed at baseline. Measurements will be registered with the digital EasyAngle Goniometer (Meloq).
Motor control of the cervical spine (craniocervical flexion test) | Baseline
  The Craniocervical flexion test (CCFT) is a clinical test of neuromotor control including the activation and endurance of the deep flexors of the cervical spine. This test involves the subject performing a "yes" like nod which is the anatomical action of the Deep Cervical flexors, against a pressure biofeedback.
  Two subscores will be used: for performance and for endurance of the deep cervical flexors.
Psychosocial headache related parameters: central sensitization by using the Central Sensitization Index (CSI). | Baseline
  The Central Sensitization Index (CSI) score ranges from 0 to 100, allowing to make the following classifications of sensitization:
  0-29 Subclinical 30-39 Mild 40-49 Moderate 50-59 Severe 60-100 Extreme
Psychosocial headache related parameters: pain catastrophizing as measured by the Pain Catastrophizing Scale (PCS) | Baseline
  The Pain Catastrophizing Scale (PCS) has 13 items, each belonging to one of three of the following subscales:
  * Rumination (item 8,9,10,11)
  * Magnification (item 6,7,13)
  * Helplessness (item 1,2,3,4,5,12) The total score of the questionnaire ranges from 0 to 52. The higher the score, the more pain catastrophizing the patient shows.
Psychosocial headache related parameters: pain coping as measured by the Pain Coping Inventory(PCI). | Baseline
  The Pain Coping Inventory (PCI) records which coping strategy is preferred by the patient. The inventory contains 6 scales which can be divided in active coping strategies (Pain Transformation, Distraction, Reducing Demands) or passive coping strategies (Retreating, Worrying, Resting).
  The higher the score per domain, the more the patients uses that type of coping.
Psychosocial headache related parameters: pain related fear as measured by the Tampa Scale of Kinesiophobia (TSK). | Baseline
  The Tampa Scale of Kinesiophobia (TSK) contains 17 items and the total score can range from 17 to 68.
  A score of more than 37 points towards kinesiophobia.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Cagnie, Prof. dr., Principal Investigator — University Ghent
Locations (1):
- University Ghent - campus UZ Ghent - Rehabilitation Sciences B3, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: No
No data will be shared outside the research team.